CLINICAL TRIAL: NCT06270888
Title: An i3+3 Phase I Hypofractionation Trial for Multiple Myeloma
Brief Title: Hypofractionation (Radiation) Trial for Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-1011
Record Dates: First submitted 2024-02-05; First posted 2024-02-21 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; radiation; bone marrow
MeSH Terms: conditions — Multiple Myeloma | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 - Dose Schedule 1 (Experimental): In this study, there will be 4 different radiation schedules, ranging from 1-10 daily treatments. Participants will be assigned to one of the dose schedules and they will know this ahead of time. The study doctor will tell each participant which study group and dose schedule they been assigned.
  For most participants, the actual time on the radiation treatment machine will be in the range of 30 to 60 minutes. The mold will be removed after the treatment. The number of treatments to each tumor will depend on which treatment group the participant is enrolled on: The longest possible treatment group would be 10 treatments in duration of about 2 weeks of treatment and the shortest possible treatment group would be 1 treatment.
  Interventions: Radiation: Radiation
- Group 2 - Dose Schedule 2 (Experimental): In this study, there will be 4 different radiation schedules, ranging from 1-10 daily treatments. Participants will be assigned to one of the dose schedules and they will know this ahead of time. The study doctor will tell each participant which study group and dose schedule they been assigned.
  For most participants, the actual time on the radiation treatment machine will be in the range of 30 to 60 minutes. The mold will be removed after the treatment. The number of treatments to each tumor will depend on which treatment group the participant is enrolled on: The longest possible treatment group would be 10 treatments in duration of about 2 weeks of treatment and the shortest possible treatment group would be 1 treatment.
  Interventions: Radiation: Radiation
- Group 3 - Dose Schedule 3 (Experimental): In this study, there will be 4 different radiation schedules, ranging from 1-10 daily treatments. Participants will be assigned to one of the dose schedules and they will know this ahead of time. The study doctor will tell each participant which study group and dose schedule they been assigned.
  For most participants, the actual time on the radiation treatment machine will be in the range of 30 to 60 minutes. The mold will be removed after the treatment. The number of treatments to each tumor will depend on which treatment group the participant is enrolled on: The longest possible treatment group would be 10 treatments in duration of about 2 weeks of treatment and the shortest possible treatment group would be 1 treatment.
  Interventions: Radiation: Radiation
- Group 4 - Dose Schedule 4 (Experimental): In this study, there will be 4 different radiation schedules, ranging from 1-10 daily treatments. Participants will be assigned to one of the dose schedules and they will know this ahead of time. The study doctor will tell each participant which study group and dose schedule they been assigned.
  For most participants, the actual time on the radiation treatment machine will be in the range of 30 to 60 minutes. The mold will be removed after the treatment. The number of treatments to each tumor will depend on which treatment group the participant is enrolled on: The longest possible treatment group would be 10 treatments in duration of about 2 weeks of treatment and the shortest possible treatment group would be 1 treatment.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Radiation given for cancer treatment. Radiation is usually an outpatient procedure completed over the course of 1-6 weeks. High-energy radiation will be delivered to a focused area of the body using a treatment machine called a linear accelerator. Unlike surgery, there are no invasive procedures other than inserting an IV during the radiation planning session. Radiation uses a mold that is customized to fit your body. This mold will be made in the radiation planning session and be used during treatment to keep you from moving. The mold is necessary for very accurate targeting of your tumor. During the procedure, the radiation therapy team will also confirm the exact location that needs to be treated using x-rays.

SUMMARY:
This study if for people who have been diagnosed with multiple myeloma and their doctors are recommending radiation to help treat it. Typically, radiation consists of 2-3 weeks of external beam radiation therapy. Doctors leading this study would like to see if a shorter radiation course (i.e., hypofractionation) for pelvic radiation is safe for multiple myeloma. Because participants in this study will receive a shortened radiation course, each daily treatment dose that is delivered would be slightly higher than normal. This higher daily dose would be delivered because the study team would like to see if higher doses of radiation are as safe given over a shorter number of days compared to 2-3 weeks. The purpose of this study is to make sure that hypofractionation is safe and effective for individuals with multiple myeloma.

DETAILED DESCRIPTION:
This study if for people who have been diagnosed with multiple myeloma and their doctors are recommending radiation to help treat it. Typically, radiation consists of 2-3 weeks of external beam radiation therapy. Doctors leading this study would like to see if a shorter radiation course (i.e., hypofractionation) for pelvic radiation is safe for multiple myeloma. Because participants in this study will receive a shortened radiation course, each daily treatment dose that is delivered would be slightly higher than normal. This higher daily dose would be delivered because the study team would like to see if higher doses of radiation are as safe given over a shorter number of days compared to 2-3 weeks. The purpose of this study is to make sure that hypofractionation is safe and effective for individuals with multiple myeloma.

In this study, there will be 4 different radiation schedules, ranging from 1-10 daily treatments. Participants in this study will be assigned to one of the dose schedules, and they will know this ahead of time. The study team will evaluate whether the shorter course of radiation is safe by monitoring and evaluating any side effects participants have that are related to the radiation schedule. As part of the research-related activities, the study team will monitor participants' side effects using assessments by their doctors; this will occur before, during, and after radiation therapy for a total of 2 years after radiation.

ELIGIBILITY:
Inclusion Criteria:

- For entry into the study, the following criteria must be met prior to dosing on Day 1. No exceptions will be granted. Eligibility criteria for this study have been carefully considered to ensure the safety of the study participants and that the results of the study can be used. It is imperative that participants fully meet all eligibility criteria.

1. Signed Written Informed Consent

   * Participants must be able to give self-consent and then sign and date an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent in accordance with local regulatory and institutional guidelines. This consent must be obtained before the performance of any protocol-related procedures that are not considered part of normal participant care.
   * Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
2. Type of Participant and Disease Characteristics

   1. General inclusion criteria:

      * Men or women ≥ 18 years of age.
      * Have clinically confirmed relapsed/refractory Multiple Myeloma with up to 5 osseous lesions that can be treated with radiation therapy (SINS score ≤ 13 or Mirels' score ≤ 9) iii) Have undergone appropriate standard of care treatment options (in the opinion of the treating investigator).

      iv) Participants must have measurable disease as defined by RECIST Version 1.1, including at least one tumor lesion that meets criteria for radiation.
      1. . 0.25 cc to 65 cc of viable tumor approximately 5 cm in maximal dimension. Tumors larger than 65 cc can be partially treated but the whole tumor should receive at least the minimal prescribed dose confirmed by the study team.

   v) Participants must have an Eastern Cooperative Oncology Group performance status that is greater than or equal to 2 vi) Adequate organ function, as defined by lab values that will be confirmed by the study doctor.
3. Age and Reproductive Status

   * Participants must be males and females ≥ 18 years of age at the time of informed consent.
   * Participants who are women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 72 hours prior to the start of study.

     c) Participants who are women must not be breastfeeding. d) Participants who are women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) and up to 5 months post last dose of study drug(s).

     e) Participants who are women of childbearing potential who are continuously not heterosexually active are exempted from contraceptive requirements but still must undergo pregnancy testing as described in this section.

     f) Participants who are males and who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) and up to 7 months post last dose of study drug(s). In addition, male participants must be willing to refrain from sperm donation during this time.

     g) Participants who are azoospermic males are exempt from contraceptive requirements.

Investigators shall counsel women of childbearing potential , and male participants who are sexually active with women of childbearing potential , on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception, which have a failure rate of < 1% when used consistently and correctly.

Exclusion Criteria:

1. Target Population

   • Participants must not have SINS (spinal instability neoplastic score) less than 13 or Mirels' score less than 9 prior to starting radiation treatment

   • Participants must not receive any concurrent anti-myeloma or systemic therapy of any form.

   • Participants who have not recovered (i.e. greater than grade 1 or at baseline) from adverse events due to a previously administered agent will be excluded. Participants may receive concurrent steroids.

   i) Note: subjects with greater than grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   ii) Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

   iii) Note: subjects with any grade alopecia are an exception to this criterion and may qualify for the study • Participants must not have had prior radiation therapy (defined as less than 10 percent of prior prescription dose) to the area planning to be treated with radiation.

   • Participants who have had prior cytotoxic chemotherapy must not receive that therapy within 2 weeks of the initiation of radiation

   • Participants who have had prior anti-cancer monoclonal antibody (mAb) or other small molecules must not receive that therapy within 7 days of the initiation of radiation

   • Participants must not have a known additional malignancy that could confuse analysis of on-study treatment. Inclusion of all study participants with more than one malignancy must be discussed and approved by the PI.
   * Participants must not have a known history of non-infectious pneumonitis that required steroids for treatment.
   * Participants must not have evidence of interstitial lung disease.
   * Participants must not have a current seizure disorder.
   * Participants must not have a history or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
   * Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
   * Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
   * If known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C is detected then patient is not eligible for treatment of liver lesions
   * Participants must not have had uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

     * Myocardial infarction or stroke/transient ischemic attack within the past 6 months
     * Uncontrolled angina within the past 3 months
     * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
     * History of other clinically significant heart disease (e.g. cardiomyopathy, congestive heart failure with New York Heart Association functional classification III to IV, pericarditis, significant pericardial effusion, or myocarditis)
     * Cardiovascular disease-related requirement for daily supplemental oxygen therapy.
   * Participants may not concomitantly use statins while on study. However, a patient using statins for over 3 months prior to study drug administration and in stable status without creatine kinase (CK) rise may be permitted to enroll.
   * Participants may not have current or history of clinically significant muscle disorders (e.g. myositis), recent unresolved muscle injury, or any condition known to elevate serum creatine kinase (CK) levels.
   * Participants must not be prisoners or be involuntarily incarcerated.
   * Participants must not be compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

   Eligibility criteria for this study have been carefully considered to ensure the safety of the study participants and that the results of the study can be used. It is imperative that participants fully meet all eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Radiation of Per Fraction | 2 years
  Maximum tolerated dose per fraction as assessed by rate of reported dose-limiting toxicities among participants.

SECONDARY OUTCOMES:
Rate of Grade 3 or Higher Adverse Events | 1 month from start of radiation
  The rate of grade 3 or higher adverse events as defined by Common Terminology Criteria for Adverse Events 5.0 that occur within 1 month from the start of radiation.
Rate of Long-Term Adverse Events | 2 Years
  The rate of long-term adverse events (after 1 month) from the end of radiation measured by an assessment of spinal osseous lesions using spinal instability neoplastic score (SINS) criteria and computed tomography (CT) imaging at first follow up.
Overall Response Rate | 2 years
  Overall response rate as assessed by clinical notes/ study records.
Progression-free Survival | 2 years
  Progression-free as assessed by clinical notes/study records.
Local Control of the treated Lesion | 2 years
  Local control of the treated lesion as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Hasan, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF